CLINICAL TRIAL: NCT05572294
Title: Mindfulness and Yoga Therapy for Acute Pain in Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Siayareh Rambally, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU-2021-0729
Record Dates: First submitted 2022-09-19; First posted 2022-10-07 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Sickle Cell Crisis; Sickle Cell Disease
Keywords: Sickle Cell Disease; Yoga Therapy; Mindfulness
MeSH Terms: conditions — Vaso-Occlusive Crises; Anemia, Sickle Cell | interventions — Mindfulness; Breathing Exercises; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness and Yoga Therapy (Experimental): Participants will have access to video-guided mindfulness interventions.
  Interventions: Behavioral: Mindfulness meditation, breathing exercises (including incentive spirometry), and yoga therapy

INTERVENTIONS:
Behavioral: Mindfulness meditation, breathing exercises (including incentive spirometry), and yoga therapy — Sickle cell patients admitted with a vaso-occlusive pain crisis over a consecutive 12-week period will be offered participation in the study. After providing informed consent, participants will have access to 4 videos containing guided mindfulness meditation, breathing exercises, and gentle yoga therapy. The videos are 5-12 minutes long and taught by a physical therapist who is also certified in yoga therapy. Participants may turn off the video at any time. Participants will have access to the videos for the duration of their hospitalization, and they may watch the videos as many times as they desire.

SUMMARY:
Patients with sickle cell disease suffer from acute and chronic pain that diminishes their quality of life. The purpose of this study is to assess the feasibility and acceptability of mindfulness meditation, breathing exercises, and gentle yoga therapy as supportive measures for the management of acute vaso-occlusive pain crises in the inpatient setting.

DETAILED DESCRIPTION:
This is a prospective single arm study of mindfulness interventions for sickle cell patients admitted with an acute vaso-occlusive pain crisis. Patients will be accrued over a consecutive 12 week period. All genotypes of sickle cell disease will be eligible for enrollment.

After providing informed consent, the patients will have access to 4 videos on their hospital room television. The videos contain guided mindfulness meditation, breathing exercises (including the use of an incentive spirometer), and gentle yoga therapy that can be performed in the supine position from a hospital bed. Videos vary in length from 5-12 minutes. Participants will have the ability to watch the videos as many times as they choose. They may also turn off the video at any time.

The primary outcome is feasibility and acceptability of the intervention. We will record objective data on how many videos are watched by each participant, as well as the percentage of each video completed. We will obtain information about the participants' perception of the intervention through a post-intervention survey and interview.

ELIGIBILITY:
Inclusion criteria:

* Patients with sickle cell disease, any genotype
* Adult patients at least 18 years of age
* English speaking
* Admitted to Clements University Hospital with an acute vaso-occlusive pain crisis

Exclusion criteria:

* Unable to follow simple instructions
* Admitted to the intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention as measured by the proportion of sickle cell patients admitted over a consecutive 12 week time period who agree to participate in the study | 12 weeks
Feasibility of the intervention as measured by the proportion of participants who accessed the mindfulness videos during their hospitalization | 12 weeks
Acceptability of the intervention as measured by the proportion of participants who found the mindfulness practices enjoyable and/or helpful | at the time of hospital discharge, up to 6 months post-intervention
  This data will be collected via a post-intervention survey and interview. The survey will contain simple questions with yes/no answer options. The interview will be conducted by a study member, either in-person or by telephone.
Acceptability of the intervention as measured by the proportion of participants who are interested in pursuing mindfulness therapies in the future | at the time of hospital discharge, up to 6 months post-intervention
  This data will be collected via a post-intervention survey and interview. The survey will contain simple questions with yes/no answer options. The interview will be conducted by a study member, either in-person or by telephone.
Participant engagement as measured by the number of mindfulness videos watched by each participant during their hospitalization | at the time of hospital discharge, up to 6 months post-intervention
Participant engagement as measured by the percentage of videos completed. A video is considered completed if the participant watches more than 85% of the video. | at the time of hospital discharge, up to 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Siayareh Rambally, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No